CLINICAL TRIAL: NCT01127386
Title: Effect of Lenalidomide (Revlimid®) in Solid Tumour Patients With Inflammatory Cancer Cachexia Syndrome on Lean Body Mass and Muscle Strength: A Multicenter, Proof-of-concept Study of Fixed Dose or CRP-response-guided Dose of Lenalidomide in Relation to New Standard Basic Cachexia Management (Receiving Placebo).
Brief Title: Lenalidomide for Lean Body Mass and Muscle Strength in Inflammatory Cancer Cachexia Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Florian Strasser, MD ABHPM (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Florian Strasser, MD ABHPM, Sponsor-Investigator, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EKSG 09/040
Record Dates: First submitted 2010-05-12; First posted 2010-05-20 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cancer Cachexia Syndrome
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fix dose lenalidomide 25mg, basic cachexia management (Experimental): dose reduction according to toxicity possible
  Interventions: Drug: Lenalidomide
- CRP-response guided lenalidomide, basic cachexia management (Experimental): start with 5mg od and increase of dosage to 10mg, 15mg or 25mg until CRP response (50% decrease)
  Interventions: Drug: Lenalidomide
- placebo (Experimental): to generate data about basic cachexia management, no direct comparator for treatment arms efficacy
  Interventions: Other: basic cachexia management (prokinetics, physical activity counselling, nutritional counselling)

INTERVENTIONS:
Drug: Lenalidomide — 25mg od, dose reduction according to toxicity
  Other Names: Revlimid
  Arms: fix dose lenalidomide 25mg, basic cachexia management
Drug: Lenalidomide — start with 5mg od and increase of dosage to 10mg, 15mg or 25mg until CRP response (50% decrease)
  Other Names: Revlimid
  Arms: CRP-response guided lenalidomide, basic cachexia management
Other: basic cachexia management (prokinetics, physical activity counselling, nutritional counselling) — twice during study
  Arms: placebo

SUMMARY:
Cancer cachexia syndrome (CCS) is frequent, causing high morbidity and mortality in affected ones. The mechanism is catabolism caused by the tumour. CRP is a surrogate marker for catabolism. There are no effective treatment options against CCS. Lenalidomide, a derivate of thalidomide, is an immunomodulatory drug (IMiD®). One of its' main effect is a decrease in inflammatory cytokines. As CCS treatment, thalidomide has shown in a randomized controlled trial to stabilize lean body mass. The effect of lenalidomide in solid tumour patients was negligible although, there might be a decrease in tumour progression. However, even if lenalidomide may be uninteresting as an anticancer treatment it might affect CCS dynamics. Respective data are currently lacking. Therefore, a dose level where an anticancer effect could be expected was chosen (group A). Relevant anti-inflammatory effect may occur below the commonly used doses to achieve tumour control, which is expected to be the main anti-cachexia effect. Therefore, a second CRP-response guided treatment arm (group B) was chosen.

Hypothesis: To test whether the response rate under new standard basic cachexia management will be at the estimated 5% and with lenalidomide (either fixed dose or CRP-guided dose) in addition to basic cachexia management at least 25%.

The primary objective of this study is to assess the efficacy of lenalidomide on lean body mass and handgrip strength in advanced solid tumour patients with inflammatory CCS.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be older than 18 years of age.
2. Tumour situation: Patients with any type of advanced (defined as locally recurrent or metastatic), incurable solid tumour.
3. Cachexia: Presence of CCS, defined as involuntary loss of weight of ≥2% in 2 months or ≥5% in 6 months, which is ongoing in the last 4 weeks, and lack of fluid retention.
4. Inflammation: CRP must be ≥ 30mg/l in the absence of any other more likely cause of increased CRP like an infection or an autoimmune disorder.
5. No simple starvation: Patients must be able to eat, defined as no severe structural barriers in the upper gastrointestinal tract and no bowel obstruction.
6. Life expectancy, physical performance: Patient must have an expected life expectancy > 3 months according to palliative performance (Pap) score and a WHO performance status (PS) ≤ 2.
7. No anti-cachexia or appetite-stimulating medications: Patients are not allowed to have corticosteroids unless for maximum 2 days per week for chemotherapy, progestin therapy, Cyclooxigenase-2 inhibitor (COX-2 inhibitor), and anabolic drugs 28 days before start of trial medication until study conclusion. Prokinetic medication, NSAR, paracetamol and novamin sulphate are allowed, if given in a fixed dose for two weeks before visit 1, and expected to be given during the whole trial period.
8. Laboratory test results: Granulocyte count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L, serum creatinine ≤ 2.0 mg/dL (177 μmol/L), creatinine clearance ClCr ≥ 50ml/min, total bilirubin ≤1.5 mg/dL (25μmol/L), and AST (SGOT)/ ALT (SGPT) ≤2 x ULN or if hepatic metastases are present ≤ 5 x ULN.
9. No other trial: Patient is not participating any other clinical intervention 28 days before start of trial medication until study conclusion.
10. Women of childbearing potential (see Annex 1): A negative pregnancy test & effective contraception are mandatory in child-bearing age.

    * A female of childbearing potential (FCBP) is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
    * A FCBP potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mU/mL within 10 to 14 days prior to and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
    * FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See (Annex 2): Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
11. Cognition: Presence of a normal level of consciousness (mandatory is a normal abbreviated screening mini-mental test or a common mini-mental ≥ 27/30; in elderly patients age ≥ 65 years or patients with low education a mini mental status of ≥25/30 points will be considered adequate).
12. Logistics: The patient is able to comply with the study schedule and procedures (including fasting for blood draws on certain visits)
13. Consent: The patient has voluntarily signed and dated the informed consent (IC), approved by the Ethics Committee (EC), prior to any study-specific procedures.

    * Will consent to the use of asprin (100mg) or low molecular weight heparin (if intolerant to aspirin) in prophylactic dose (e.g. Fragmin 2500U sc od).
    * Study participant agrees to be registered in the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.(Appendix 18)

Exclusion Criteria:

1. Untreated secondary causes of cachexia (oral thrush, nausea, vomiting, constipation, diarrhoea, pain VAS>3, depression, dyspnoea)
2. CTCAEv3.0 ≥ grade 2 due to anticancer treatment (chemotherapy, radiotherapy or surgery)
3. Any psychiatric disorder, alcohol and illicit drug abuse or language problem that would prevent the patient from filling in the questionnaires adequately or attend study visits according to protocol.
4. Parenteral nutrition
5. Presence of dysthyreosis, defined as TSH beyond normal ranges
6. Presence of long QT syndrome or QTc > 450ms or under treatment with a QT prolonging drug
7. Presence of lactose intolerance
8. Diabetes mellitus with secondary organ dysfunction (coronary heart disease, previous stroke, renal insufficiency)
9. Patients with cerebral metastases or prophylactic whole brain irradiation for possible cerebral metastases.
10. Known hypersensitivity to thalidomide or a history of development of erythema nodosum due to thalidomide or similar drugs.
11. Any prior use of lenalidomide
12. Known infection with HIV, hepatitis B or C
13. Patients with known myeloid malignancy or tumours having bone marrow involvement.
14. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
15. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent (IC) form.
16. Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-03; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Lean Body Mass | after 8 weeks treatment
and Handgrip Strength | after 8 weeks treatment

SECONDARY OUTCOMES:
SAEs | for 12 weeks
nutritional intake | after 8 weeks of treatment
physical functioning | after 8 weeks of treatment
inflammation | for 8 weeks
eating related symptoms (FAACT) | after 8 weeks of treatment
tumour dynamics (CT) | after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland